CLINICAL TRIAL: NCT00275015
Title: Pivotal Study for High Dose Therapy and Autologous Stem Cell Transplantation in Early Stages of CLL
Brief Title: Cyclophosphamide and Total Body Irradiation in Treating Patients Who Are Undergoing an Autologous Peripheral Stem Cell Transplant For Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL3; EU-20553
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Carmustine; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; fludarabine phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

ARMS (1):
- High dose therapy + autologous PBSCT (Experimental): 1. Cytoreductive treatment: (preferentially) FC (2-4 cycles)
  2. Mobilization: Dexa-BEAM + G-CSF (1-2 cycles)
  3. Myeloablation:
     fractionated TBI (e.g. 6x2Gy) + Cyclophosphamide (2 x 60 mg/kg; d -4 to -3)
  4. autologous peripheral blood stem cell transplantation (PBSCT) (d 0)
  Interventions: Biological: filgrastim; Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: etoposide; Drug: fludarabine phosphate; Drug: melphalan; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: fludarabine phosphate
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy before a peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy or radiation therapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy.

PURPOSE: This phase II trial is studying how well giving cyclophosphamide together with total-body irradiation works in treating patients who are undergoing an peripheral stem cell transplant for chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of autologous peripheral blood stem cell transplantation in patients with chronic lymphocytic leukemia treated with cyclophosphamide and total-body irradiation.

Secondary

* Determine the safety, feasibility, and efficacy of combination therapy comprising dexamethasone, carmustine, cytarabine, etoposide, and melphalan (Dexa-BEAM) and filgrastim (G-CSF) mobilization in patients treated with this regimen.
* Determine the efficacy of ex-vivo graft purging in patients treated with this regimen.
* Determine the incidence of complete clinical and molecular remissions in patients treated with this regimen.
* Determine the progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter, open-label, nonrandomized study.

* Cytoreductive treatment: Patients undergo 2-4 courses of cytoreductive treatment, preferably following the fludarabine and cyclophosphamide (FC) protocol.
* Stem cell mobilization: Patients achieving a complete remission (CR) or partial remission (PR) and stable blood counts undergo stem cell mobilization comprising dexamethasone, carmustine, cytarabine, etoposide, melphalan (Dexa-BEAM), and filgrastim (G-CSF). Patients with an adequate number of mobilized cells undergo stem cell collection. Patients with CR or very good PR proceed to myeloablative therapy.
* Myeloablative therapy: Patients undergo total-body irradiation on day -4 and receive cyclophosphamide IV on days -4 and -3.
* Autologous peripheral blood stem cell transplantation (PBSCT): Patients undergo autologous PBSCT on day 0.

After completion of study, patients are followed periodically.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with chronic lymphocytic leukemia, meeting 1 of the following criteria:

  * Binet stage B or C disease
  * Binet stage A disease and at high risk for disease progression, defined as the following:

    * Non-nodular marrow infiltration or lymphocyte doubling time < 12 months
    * Thymidine kinase > 7.0 U/L or ß-2-microglobulin > 3.5 mg/L
* Polymerase chain reaction-amplifiable clonal CDRIII rearrangement of the IgV_H

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* No concurrent disease resulting in major organ dysfunction

PRIOR CONCURRENT THERAPY:

* No prior combination therapy comprising melphalan, dexamethasone, carmustine, cytarabine, and etoposide (DEXA-Beam)
* No more than 1 prior chemotherapy regimen
* No prior chemotherapy regimen longer than 6 months in duration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 1998-01; Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety of autologous peripheral stem cell transplantation (PBSCT) as measured by a treatment-related mortality of < 5% at 12 months following transplant
Feasibility of PBSCT as measured by > 50% of included patients proceeding to transplant

SECONDARY OUTCOMES:
Safety of mobilization comprising dexamethasone, carmustine, cytarabine, etoposide, and melphalan (Dexa-BEAM) as measured by a treatment-related mortality of < 5% before transplant phase
Efficacy of Dexa-BEAM mobilization as measured by the amount of CD34+ cells > 4x10e6/kg at harvest
Complete clinical remissions by NIH criteria at 3 months following transplant
Molecular remissions by CDR3 PCR at 3 months following transplant
Progression-free survival by NIH criteria at 5 years from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dreger, Study Chair — Universitaets-Kinderklinik Heidelberg
Locations (53):
- Austria (2):
  - Allg. Krankenhaus der Stadt Wien Universitaets-Kinderklinik, Vienna
  - Hanuschkrankenhaus, Vienna
- Germany (51):
  - Humaine - Clinic, Bad Saarow
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Praxis Dres. F.& G. Doering, Bremen
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Michael Schaefers und Partner, Duisburg
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Onkologische Schwerpunkt Praxis, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Malteser Krankenhaus, Flensburg
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - Universitätsklinikum Göttingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Asklepios Klinik St. Georg, Hamburg
  - St. Marien-Hospital Hamm - Klinik Knappenstrasse, Hamm
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Gemeinschaftspraxis fuer Haematologie, Onkologie und Infektiologie, Karlsruhe
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Staedtisches Krankenhaus Kiel, Kiel
  - University Leipzig Clinic of Internal Medicine, Leipzig
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Sana Kliniken Luebeck, Lübeck
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Universitatsklinik Mainz, Mainz
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universitaet Muenchen - Innenstadt Campus, Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - University of Muenster, Münster
  - Internistische Praxis - Neuss, Neuss
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Klinikum Ernst Von Bergmann, Potsdam
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Buergerhospital Stuttgart, Stuttgart
  - Internistische Praxis - Trier, Trier
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - University Wurzburg, Würzburg

REFERENCES:
- [Result] Dreger P, Dohner H, McClanahan F, Busch R, Ritgen M, Greinix H, Fink AM, Knauf W, Stadler M, Pfreundschuh M, Duhrsen U, Brittinger G, Hensel M, Schetelig J, Winkler D, Buhler A, Kneba M, Schmitz N, Hallek M, Stilgenbauer S; German CLL Study Group. Early autologous stem cell transplantation for chronic lymphocytic leukemia: long-term follow-up of the German CLL Study Group CLL3 trial. Blood. 2012 May 24;119(21):4851-9. doi: 10.1182/blood-2011-09-378505. Epub 2012 Apr 5. PMID 22490331